CLINICAL TRIAL: NCT02170259
Title: Efficacy of Manual Therapy for the Treatment of Tension-type Headache in Patients With Anxiety and Depressive Disorders. A Randomized Controlled Clinical Trial
Brief Title: Manual Therapy for Tension Headache With Psychological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhDr, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UVtensiontype
Record Dates: First submitted 2014-06-03; First posted 2014-06-23 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Tension-type Headache
Keywords: Tension-type headache; Depression; Anxiety; Manual therapy; Spinal manipulation; Patients diagnosed with tension-type headache
MeSH Terms: conditions — Tension-Type Headache; Depression; Anxiety Disorders | interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- suboccipital technique (Experimental): The suboccipital technique (ST) aims to release the spasm of the muscles affected in tension-type headaches and in general of suboccipital soft tissues, as they are responsible for the mobility dysfunction of the occiput-atlas-axis joint; this releases the facial restriction of this region.
  Interventions: Other: The suboccipital technique
- The articulatory technique (Experimental): - The articulatory technique (AT) was administered to correct and restore the mobility of joints between occiput, atlas and axis - correcting a global joint dysfunction. This technique was performed in supine position, in the same manner as the preceding technique, bilaterally and in two phases.
  Interventions: Other: The articulatory technique
- Combined treatment (Experimental): Combined treatment (ST and AT). Combination treatment consisted of the application of the two preceding treatments in the same sequence: first, treatment with ST and then AT.
  Interventions: Other: Combined treatment
- Control group (No Intervention): Control group. The control group was not applied a treatment technique

INTERVENTIONS:
Other: The suboccipital technique — The suboccipital technique (ST) aims to release the spasm of the muscles affected in tension-type headaches and in general of suboccipital soft tissues, as they are responsible for the mobility dysfunction of the occiput-atlas-axis joint; this releases the facial restriction of this region. Patients lied on the stretcher, in supine position, with their occiput resting against the physiotherapist's hands. Fingertips slide until contacting the posterior arch of atlas so that it "hangs" from the fingers. A deep and progressive pressure is applied, perpendicularly to muscle fibers, until the therapist perceives that muscle tone decreases. Approximate duration of ST is 10 minutes and it is performed with patients' eyes closed because of the connection between craniocervical muscle tone and eye movements
  Arms: suboccipital technique
Other: The articulatory technique — The articulatory technique (AT) was administered to correct and restore the mobility of joints between occiput, atlas and axis - correcting a global joint dysfunction. This technique was performed in supine position, in the same manner as the preceding technique, bilaterally and in two phases. First, a gentle head decompression is applied, followed by small circumduction searching for the joint barrier in rotation through selective tension. Second, the manipulation is performed by a cranial rotation towards the same side as the circumduction and around a vertical axis passing through the axis, without cervical flexion or extension and very little bending
  Arms: The articulatory technique
Other: Combined treatment — Combined treatment (ST and AT). Combination treatment consisted of the application of the two preceding treatments in the same sequence: first, treatment with ST and then AT, thereafter maintaining the resting position for five minutes
  Arms: Combined treatment

SUMMARY:
Introduction. Tension-type headache is a highly prevalent disorder with a significant socio-economic impact, affecting psychological aspects. This study aims to assess aspects pertaining to anxiety, depression, headache frequency and pain intensity.

Subjects and methods. A clinical trial was conducted on 84 participants suffering from tension-type headache, divided into 4 groups, the mean age being 39.76 years (SD 11.38). The first group received suboccipital soft tissue treatment (ST); the second group was treated with articulatory technique (AT); the third group was applied a combination of both techniques (ST and AT) and a forth group which served as control group. Treatment sessions were administered during four weeks, with a post-treatment assessment, and follow-up after one month. The investigators conducted Repeated measures Analysis of Covariance (RM-MANCOVA) to evaluate the effect of treatment on between and within-subject conditions and their interaction on reported depression, anxiety, and headache pain frequency and intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in this study had been diagnosed in primary healthcare centers with frequent episodic tension-type headache (ETTH) or chronic tension-type headache (CTTH) as described by the International Headache Society (IHS). Participants presented pericranial tenderness evolving over a period greater than six months and all were pharmacologically stable.

Exclusion Criteria:

* Exclusion criteria covered patients with secondary headache suffering from photophobia or phonophobia, nausea or vomiting, cases of headache aggravated by head movements, musculoskeletal disorders, previous neck trauma, vertigo, dizziness, arterial hypertension, arthritis or advanced degenerative osteoarthritis, patients with heart devices, excessive emotional tension, neurological disorders, radiological alterations, pregnancy and a positive vertebral artery test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Frequency of TTH at week 4 and at week 8 | Baseline, week 4, and week 8
  During the study, all subjects completed a weekly register of headaches.
Change from baseline in Intensity of TTH at week 4 and at week 8 | Basline, week 4 and week 8
  During the study, all subjects completed a weekly register of headaches, recording on a daily basis their intensity, using the Visual Analogue Scale (VAS), which measures pain intensity in a 0-10 scale (0=no pain, 10=the most severe pain).

SECONDARY OUTCOMES:
Anxiety | All patients were assessed under the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks).
  Anxiety was assessed with the State-Trait Anxiety Inventory (STAI-SA and STAI-TA). Scores range from 0 to a maximum of 60 points; scoring above the 50th percentile indicates the presence of anxiety. For men, this percentile correlates with a score of 19 points, both for STAI-state and STAI-trait. For women, scores over 21 for STAI-state and 24 for STAI-trait determine this level.
Depression | All patients were assessed under the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks).
  Depression, assessed with the Beck Depression Inventory (BDI) , which consists of 21 items with 4 possible answers each; it is intended to assess the severity of depression. It was adapted into Spanish and validated by Conde and Useros, showing very good

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma v. Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Result] Penacoba-Puente C, Fernandez-de-Las-Penas C, Gonzalez-Gutierrez JL, Miangolarra-Page JC, Pareja JA. Interaction between anxiety, depression, quality of life and clinical parameters in chronic tension-type headache. Eur J Pain. 2008 Oct;12(7):886-94. doi: 10.1016/j.ejpain.2007.12.016. Epub 2008 Mar 10. PMID 18331805